CLINICAL TRIAL: NCT01850355
Title: An Open-label Trial of Buspirone for the Treatment of Anxiety in Youth With Autism Spectrum Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Gagan Joshi, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013-P-000661
Record Dates: First submitted 2013-04-22; First posted 2013-05-09 (Estimated); Results first posted 2025-02-25 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Autism Spectrum Disorders; Anxiety
Keywords: Autism Spectrum Disorders; Anxiety; Children; Adolescents; Buspar; Buspirone; Pervasive Developmental Disorders
MeSH Terms: conditions — Autism Spectrum Disorder; Anxiety Disorders; Child Development Disorders, Pervasive | interventions — Buspirone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Buspirone (Experimental): Buspirone administered in tablets twice daily titrated to a maximum daily dose of 60mg for 8 weeks.
  Interventions: Drug: Buspirone

INTERVENTIONS:
Drug: Buspirone — Children with autism spectrum disorders will receive buspirone treatment for eight weeks. Buspirone will be titrated to the maximum daily dose during the first four weeks of the trial (dose titration phase). Week 4 onwards, subjects will be maintained on maximum achieved dose until the end of the trial (dose maintenance pahe). During the titration phase, total dose will be increased by 10mg at each visit and by 5mg on the 4th day after each visit.

SUMMARY:
The main objective of this exploratory 8-week pilot study is to evaluate the safety and efficacy of buspirone for the treatment of anxiety in youth (ages 6-17 years) with autism spectrum disorders. The study results will be used to generate hypothesis for a larger randomized controlled clinical trials with explicit hypotheses and sufficient statistical power.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants between 6 and 17 years of age
* Fulfills diagnosis of autism spectrum disorders by meeting DSM-IV-TR PDD diagnostic criteria of autistic disorder, Asperger's disorder, or PDD-NOS as established by clinical diagnostic interview
* Participants with a score of ≥13 on the Pediatric Anxiety Rating Scale (PARS)
* Participants with a score of ≥60 or more on the Anxiety/Depression subscale of CBCL and CGI-Anxiety severity of ≥ 4
* Subjects can be on psychotropic drugs if they have been on the medication for at least 4 weeks prior to initiating trial treatment and if they are stable, provided the medication is not listed in the Concomitant Medications section of the protocol.
* Subjects with disruptive behavior disorders, mood, or psychosis will be allowed to participate in the study provided they do not meet any exclusionary criteria

Exclusion Criteria:

* I.Q. < 70
* DSM-IV-TR PDD diagnoses of Rett's disorder, and childhood disintegrative disorder
* History of active seizure disorder (EEG suggestive of seizure activity and/or history of seizure in last 1 month)
* Subjects with a medical condition or treatment that will either jeopardize subject safety or affect the scientific merit of the study, including:
* Pregnant or nursing females
* Organic brain disorders
* Uncorrected hypothyroidism or hyperthyroidism
* Clinically significant abnormalities on ECG (e.g., QT prolongation, arrhythmia)
* History of renal or hepatic impairment
* Clinically unstable psychiatric conditions or judged to be at serious suicidal risk
* Current diagnosis of schizophrenia
* History of substance use (except nicotine or caffeine) within past 3 months or urine drug screen positive for substances of abuse
* Current treatment with medication with primary central nervous system activity (as specified in the Concomitant Medication section of the protocol)
* A non-responder or history of intolerance to buspirone, after treatment at an adequate dose and duration as determined by the clinician
* Subjects currently taking monoamine oxidase inhibitors (MAOI) and/or CYP3A4 inducers or inhibitors including nefazodone, diltiazem, verapamil, erythromaycin, itraconazole, or rifampin.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 9 (Actual)
Dates: Start 2013-07 (Actual); Primary Completion 2024-12 (Actual); Study Completion 2024-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gagan Joshi, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Participants Ages 6-17: Participants ages 6-17 with autism spectrum disorders and anxiety enrolled to receive treatment with buspirone
Period: Overall Study
Arm/Group | Participants Ages 6-17
Started | 9
Completed | 6
Not Completed | 3

BASELINE CHARACTERISTICS:
Arm/Group | Participants Ages 6-17
Number analyzed (Participants) | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 9
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.7 (2.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 9
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 8
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 9

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Pediatric Anxiety Rating Scale (PARS)
Description: The PARS is a clinician-rated scale to be used with parents and children. It consists of 57 items and has two sections: a symptom checklist (first 50 items) and severity items (last 7 items). The symptom checklist is used to determine the child's repertoire of symptoms during the past week. The 7 severity items are used to determine severity of symptoms and the PARS total score. The total score for the PARS is derived by summing the 7 severity items; total score ranges from 0 to 35, where higher scores indicate greater severity. The outcome reported reflects the change from baseline in PARS scores. When examining change from baseline, negative scores represent improvement (i.e., decrease in severity from baseline).
Time Frame: Baseline to week 8
Population: Participants who were exposed to study medication for at least two weeks. One participant was not included because they withdrew consent prior to starting treatment.
Measure: Mean (Standard Deviation); unit: change in scale score
Groups:
- Participants Ages 6-17: Participants ages 6-17 enrolled to receive buspirone treatment
Arm/Group | Participants Ages 6-17
Number analyzed (Participants) | 8
change in scale score | -10.3 (6.4)

2. Primary Outcome: Clinician-rated Clinical Global Impression-Anxiety-Improvement (CGI-Anxiety-I) Scores of Improved or Very Much Improved at Study Endpoint
Description: The CGI-Anxiety-I is a clinician rated measure of anxiety improvement. Improvement scores range from 1 (very much improved) to 7 (very much worse). This outcome reports the number of participants who scored ≤2 (improved or very much) at study endpoint.
Time Frame: Week 8 (study endpoint)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Participants Ages 6-17
Number analyzed (Participants) | 8
participants | 4

3. Primary Outcome: Treatment Responder
Description: Treatment responder is defined by a Clinician-rated Clinical Global Impression-Anxiety-Improvement (CGI-Anxiety-I) score ≤ 2 (improved or very much improved) and a ≥30% reduction on the Pediatric Anxiety Rating Scale (PARS) from baseline.
Time Frame: Week 8 (study endpoint)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Participants Ages 6-17
Number analyzed (Participants) | 8
participants | 4

ADVERSE EVENTS:
Time Frame: 8 weeks (from baseline to end of study)
Description: One participant withdrew consent prior to starting treatment and is not included in the adverse event reporting.
Arm/Group | Participants Ages 6-17
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 8/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Participants Ages 6-17 (N=8)
Headache (General disorders) | 3 (5)
Irritability (Psychiatric disorders) | 3 (3)
Insomnia (Nervous system disorders) | 2 (3)
Nausea (Gastrointestinal disorders) | 1 (2)
Dizziness (General disorders) | 1 (2)
Drowsiness (General disorders) | 1 (2)
Fatigue (General disorders) | 1 (2)
Palpitations (Cardiac disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-12-14): https://cdn.clinicaltrials.gov/large-docs/55/NCT01850355/Prot_SAP_000.pdf